CLINICAL TRIAL: NCT04041245
Title: A Study on the Metabolic Characteristics of Meridian Phenomenon for the Heart and Lung Meridians Based on Patients With Stable Angina Pectoris
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhejiang Chinese Medical University (Other Government)
Collaborators: The Third Affiliated hospital of Zhejiang Chinese Medical University (Other); The First Affiliated Hospital of Zhejiang Chinese Medical University (Other)
Responsible Party: Principal Investigator, Jianqiao Fang, President, Zhejiang Chinese Medical University
Other Study IDs: 2019ZY002-MERIDIAN
Record Dates: First submitted 2019-07-26; First posted 2019-08-01 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2019-08

CONDITIONS: Chronic Stable Angina Pectoris
Keywords: meridians; acupuncture; chronic stable angina pectoris; meridian phenomenon; near infrared spectroscopy
MeSH Terms: interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CSAP group: This group will include 40 patients with chronic stable angina pectoris (CSAP).
  Interventions: Device: Near infrared spectroscopy
- Healthy group: This group will include 40 healthy volunteers.
  Interventions: Device: Near infrared spectroscopy

INTERVENTIONS:
Device: Near infrared spectroscopy — Near infrared spectroscopy will be adopted to assess the microcirculatory characteristics of meridian phenomenon for participants in the two groups.
  1. Experimental device: a four-channel INVOS 5100C Oximeter (Somanetics Corp., Troy, USA)
  2. Experimental process: The participants will be allowed to stabilize for 15 minutes in a supine position in the experimental room before formal examination.
     They are asked to keep silent, breathe normally and avoid movement of limbs during the whole measuring period. After ripping the transparent adhesive tape on the probe, the probes will be left at 4 measuring sites. Regional oxygen saturation (rSO2) will be recorded for 5 minutes.
  3. Measurement sites: Shenmen (HT7) and Shaohai (HT3) of the Heart meridian, Taiyuan(LU9) and Chize (LU5) of the Lung meridian.

SUMMARY:
Although some important progresses were made in the field of the meridian research, no breakthroughs have been achieved. Besides,there are some problems in meridian researches. Particularly, previous research of meridian phenomenon involved lots of subjective elements and outcomes.Researches that use modern scientific techniques to investigate the biological characteristics of meridian phenomenon are urgently needed. Therefore, this study is designed to assess the metabolic characteristics of meridian phenomenon for the Heart and Lung meridians by using near infrared spectroscopy. Thus, the biological characteristics of meridian phenomenon could be presented objectively in a scientific methodology.

DETAILED DESCRIPTION:
This study will include 40 patients diagnosed with chronic stable angina pectoris (CSAP) and 40 healthy volunteers. Near infrared spectroscopy will be adopted to assess the metabolic characteristics of meridian phenomenon for Heart and Lung meridians in the physiology/pathological state. In addition, by comparing the metabolic characteristics in the acupoints along the Heart and Lung meridians, the relative specificity of the two meridians will also be investigated.

Primary outcomes will be regional oxygen saturation (rSO2). Furthermore, this study will build standardized techniques and schemes for detecting the metabolic characteristics of meridian phenomenon for Heart and Lung. The results of this study could also provide scientific foundation for traditional meridian theories.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for CSAP

1. Patients should meet the diagnostic criteria of coronary heart disease, which includes the following items: 1)confirmed old myocardial infarction (MI), or a history of percutaneous coronary intervention(PCI), or coronary artery bypass grafting; 2)50% or more luminal stenosis in at least one coronary artery or major branch segment confirmed by coronary angiogram or CT angiography; 3) myocardial ischemia indicted by exercise stress radionuclide myocardial imaging; 4) treadmill exercise testing is positive (for male patients);
2. Patients should meet the diagnostic criteria of CSAP and the Canadian Cardiovascular Society(CCS) classification for CSAP is level II or III;
3. The medical history of angina pectoris ≥3 months, with at least 2 episodes per week in the last month;
4. 35 ≤ age ≤65 years, male or female;
5. Patients have clear consciousness and could communicate with others normally;
6. Patients could understand the full study protocol and have high adherence. Written informed consent is signed by themselves or their lineal kin.

Inclusion criteria for health volunteers

1. Healthy volunteers who could provide a recent (in the past 3 month) medical examination report to confirm they have not any cardiovascular, respiratory, digestive, urinary, hematological, endocrine and neurological disease;
2. 35 ≤ age ≤65 years, male or female;
3. Participants have clear consciousness and could communicate with others normally;
4. Participants could understand the full study protocol and have high adherence .Written informed consent is signed by themselves or their lineal kin.

Exclusion Criteria:

Exclusion criteria for CSAP

1. Patients with acute coronary syndrome (including acute myocardial infarction and unstable angina) and severe arrhythmias (such as severe atrioventricular block, ventricular tachycardia, supraventricular tachycardia, frequent premature beats and premature ventricular contraction);
2. Patients' chest pain is caused by valvular heart disease, hypertrophic cardiomyopathy and dilated cardiomyopathy;
3. Patients' chest pain is caused by non-cardiac disease (such as severe neurosis, climacteric syndrome, cervical spondylosis, and esophageal/pulmonary/chest wall lesions);
4. Patients have concomitant conditions of lung diseases, such as COPD;
5. Patients have serious concomitant conditions and and fail to treat them effectively, such as diseases of the digestive, urinary, respiratory, hematological and nervous system;
6. Patients have mental illness, severe depression, alcohol dependence or history of drug abuse;
7. Pregnant or lactating patients;
8. Patients are participating in other trials.

Exclusion criteria of health volunteers

1. Participants have sudden severe diseases during the trial, such as cardiovascular diseases, liver diseases, kidney diseases, urinary diseases and hematological diseases.
2. Participants have mental illness, severe depression, alcohol dependence or history of drug abuse;
3. Pregnant or lactating participants ;
4. Participants are participating in other trials.

Ages: 35 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 40 patients with chronic stable angina pectoris (CSAP) and 40 healthy volunteer.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Regional oxygen saturation (rSO2) | 5 minutes
  Regional oxygen saturation could reflect the metabolic characteristics of meridians phenomenon.

CONTACTS AND LOCATIONS:
Overall Officials: Jianqiao Fang, Ph.D, Principal Investigator — Zhejiang Chinese Medical University
Locations (1):
- the Third affiliated hospital of Zhejiang Chinese Medical university, Hanzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Litscher G, Wang L. [Cerebral near infrared spectroscopy and acupuncture--results of a pilot study]. Biomed Tech (Berl). 2000 Jul-Aug;45(7-8):215-8. doi: 10.1515/bmte.2000.45.7-8.215. German. PMID 10975151
- [Background] Raith W, Pichler G, Sapetschnig I, Avian A, Sommer C, Baik N, Koestenberger M, Schmolzer GM, Urlesberger B. Near-infrared spectroscopy for objectifying cerebral effects of laser acupuncture in term and preterm neonates. Evid Based Complement Alternat Med. 2013;2013:346852. doi: 10.1155/2013/346852. Epub 2013 May 15. PMID 23762122
- [Background] Litscher G, Wang L, Huber E. [Changes in cerebral near infrared spectroscopy parameters during manual acupuncture needle stimulation]. Biomed Tech (Berl). 2002 Apr;47(4):76-9. doi: 10.1515/bmte.2002.47.4.76. German. PMID 12051136
- [Background] Takamoto K, Hori E, Urakawa S, Sakai S, Ishikawa A, Kohno S, Ono T, Nishijo H. Cerebral hemodynamic responses induced by specific acupuncture sensations during needling at trigger points: a near-infrared spectroscopic study. Brain Topogr. 2010 Sep;23(3):279-91. doi: 10.1007/s10548-010-0148-8. Epub 2010 May 26. PMID 20502956
- [Background] Litscher G, Wang L, Schwarz G, Schikora D. [Increases of intracranial pressure and changes of blood flow velocity due to acupressure, needle and laser needle acupuncture?]. Forsch Komplementarmed Klass Naturheilkd. 2005 Aug;12(4):190-5. doi: 10.1159/000087044. Epub 2005 Aug 29. German. PMID 16137980
- [Background] Litscher G, Schwarz G, Sandner-Kiesling A, Hadolt I, Eger E. Effects of acupuncture on the oxygenation of cerebral tissue. Neurol Res. 1998;20 Suppl 1:S28-32. doi: 10.1080/01616412.1998.11740605. PMID 9584920
- [Background] Ohkubo M, Hamaoka T, Niwayama M, Murase N, Osada T, Kime R, Kurosawa Y, Sakamoto A, Katsumura T. Local increase in trapezius muscle oxygenation during and after acupuncture. Dyn Med. 2009 Mar 16;8:2. doi: 10.1186/1476-5918-8-2. PMID 19291290
- [Background] Litscher G, Ofner M, He W, Wang L, Gaischek I. Acupressure at the Meridian Acupoint Xiyangguan (GB33) Influences Near-Infrared Spectroscopic Parameters (Regional Oxygen Saturation) in Deeper Tissue of the Knee in Healthy Volunteers. Evid Based Complement Alternat Med. 2013;2013:370341. doi: 10.1155/2013/370341. Epub 2013 Feb 7. PMID 23476689
- [Background] Banzer W, Hubscher M, Seib M, Vogt L. Short-time effects of laser needle stimulation on the peripheral microcirculation assessed by laser Doppler spectroscopy and near-infrared spectroscopy. Photomed Laser Surg. 2006 Oct;24(5):575-80. doi: 10.1089/pho.2006.24.575. PMID 17069486
- [Background] Jimbo S, Atsuta Y, Kobayashi T, Matsuno T. Effects of dry needling at tender points for neck pain (Japanese: katakori): near-infrared spectroscopy for monitoring muscular oxygenation of the trapezius. J Orthop Sci. 2008 Mar;13(2):101-6. doi: 10.1007/s00776-007-1209-z. Epub 2008 Apr 8. PMID 18392913
- [Background] Murkin JM, Arango M. Near-infrared spectroscopy as an index of brain and tissue oxygenation. Br J Anaesth. 2009 Dec;103 Suppl 1:i3-13. doi: 10.1093/bja/aep299. PMID 20007987
- See also: Near-infrared spectroscopy for objectifying cerebral effects of needle and laserneedle acupuncture — https://www.researchgate.net/publication/242230245_Near-Infrared_Spectroscopy_For_Objectifying_Cerebral_Effects_Of_Needle_And_Laserneedle_Acupuncture

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-03-25): https://cdn.clinicaltrials.gov/large-docs/45/NCT04041245/Prot_SAP_000.pdf
  • Informed Consent Form (2019-03-25): https://cdn.clinicaltrials.gov/large-docs/45/NCT04041245/ICF_001.pdf